CLINICAL TRIAL: NCT05699018
Title: Screening in Primary Care of Advanced Liver Fibrosis in NAFLD And/or Alcoholic Patients
Acronym: SOPRANO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022-A02148-35
Record Dates: First submitted 2022-12-28; First posted 2023-01-26 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Alcoholic Liver Disease (ALD); Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases, Alcoholic; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: The SOPRANO study is a multicenter prospective comparative diagnostic study . Evaluation of a simple blood test (e-LIFT) for the diagnosis of advanced liver fibrosis.
  Reference for advanced liver diagnosis : composite criteria :
  * Elastometry between 8 kPa and 14.9 kPa and histologic evaluation of fibrosis ≥ F3 (NASH CRN ) OR
  * Elastometry ≥ 15 kPa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Test: e-LIFT (Other): only one arm because diagnostic study evaluating blood test using elastometry and liver biopsy as reference
  Interventions: Diagnostic Test: eLIFT

INTERVENTIONS:
Diagnostic Test: eLIFT — Diagnostic procedure: elastography devices, blood tests (e-LIFT + Fibrometer), liver biopsy if necessary (elastometry ≥ 8 kPa and < 15 kPa)

SUMMARY:
The primary objective of the SOPRANO study is to compare two blood fibrosis tests, the eLIFT and the FibroMeter, for the screening of advanced liver fibrosis in patients with NAFLD and/or ALD from primary care centers.

DETAILED DESCRIPTION:
Chronic liver diseases (CLD) are responsible for 17 000 deaths each year in France (cirrhosis: 8 000, liver cancer: 9 000). Non-alcoholic fatty liver disease (NAFLD) and alcoholic liver disease (ALD) are the two main causes of CLD in France, affecting respectively 25% and 12% of the adult general population. A subset of these patients develops advanced liver fibrosis (ALF), which requires referral to the specialist for specific evaluation and management to avoid the occurrence of cirrhosis and its life-threatening complications. General practitioners (GPs) are the first-line physicians in front of the large population of NAFLD and/or ALD patients. It is very difficult for GPs to identify the patients who develop ALF and require referral to the specialist, as their physical examination, usual biology and ultrasonography remain normal.

The non-invasive diagnosis of liver fibrosis is now available with elastography devices and blood tests. Elastography is a very accurate method but it is available only in few specialised centers. Specialised blood tests are available to all physicians, but they are quite expensive and not reimbursed with therefore limited use in clinical practice. Consequently, liver fibrosis remains unevaluated in most patients with NAFLD and/or ALD, which explains why a lot are too late diagnosed at the stage of cirrhosis complications with poor short-term survival.

The eLIFT isa new blood fibrosis test specifically dedicated for GPs with simple parameters and easy "by head" calculation. The simple eLIFT was compared with the specialised blood test FibroMeter for the diagnosis of ALF in an cohort of 1024 biopsy-proven NAFLD and/or ALD patients. eLIFT was little less accurate than FibroMeter (AUROC: 0.78 vs 0.81). Using the recommended cut-offs (eLIFT ≥8, FibroMeter ≥0.46), eLIFT was more sensitive than FibroMeter (86% vs 77%), whereas FibroMeter was highly more specific (71% vs 51%). These results position eLIFT and FibroMeter as interesting tools for the screening of ALF in large populations.

As the preliminary results come from very selected patients, i.e. patients from tertiary centers who underwent a liver biopsy, it's necessary nox to evaluate in the real condition of primary care setting whether the use of eLIFT or FibroMeter will help GPs to screen ALF in their asymptomatic NAFLD and ALD patients.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD and/or ALD patient defined by at least 1 of the following criteria:

  * Excessive alcohol consumption: higher than 210 g / week (men), or 140 g / week (women)
  * Type 2 diabetes
  * at least 2 metabolic factors among BMI higher than or equal to 25 kg / m 2; Elevated blood pressure (antihypertensive drug, or systolic blood pressure higher than or equal to 130mmHg, or diastolic blood pressure higher than or equal to 85mmHg), Dyslipidemia (lipid-lowering drug, or HDL cholesterol lower to 40mg/dl (men) / 50mg/dl (women), or triglycerides higher than or equal to150mg/dl); Hyperferritinemia (higher than upper limit of normal from the laboratory)
  * Bright liver at ultrasonography without steatosis-inducing drug(systemic corticosteroids, tamoxifen, amiodarone, methotrexate)

Following a protocol amendment, the 3 last investigating primary care centres will include NAFLD and/or ALD patients according to these updated criteria:

* Excessive alcohol consumption: >210 g/week in men or >140 g/week in women,
* AND/OR type 2 diabetes treated with insulin and/or at least two other anti-diabetic treatments,
* AND with the following stratification:

  40% with excessive alcohol consumption 40% with type 2 diabetes treated with insulin and/or at least two other anti-diabetic treatments 20% with both conditions (excessive alcohol consumption, AND type 2 diabetes treated with insulin and/or at least two other anti-diabetic treatments)
* Patient's agreement to have a blood sample collected in a local laboratory participating in the study
* Subjects covered by or having the rights to medical care assurance
* Written informed consent obtained from subject

Exclusion Criteria:

* Already ongoing specialized follow-up for a chronic liver disease
* Altered health status with poor short-term prognosis, not compatible with a screening procedure
* Decompensated cirrhosis (hepatic encephalopathy, jaundice, ascites, variceal bleeding, hepatorenal syndrome)
* Acute infection
* Pregnancy, breastfeeding
* Persons in detention by judicial or administrative decision
* Person admitted to a health or social establishment for purposes other than research
* Person subject to a legal protection measure
* Person unable to express consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1788 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the eLIFT test for advanced liver fibrosis | 1 day
  Rate of patients with advanced liver fibrosis correctly identified by the eLIFT test
Sensitivity of the Fibrometer test for advanced liver fibrosis | 1 day
  Rate of patients with advanced liver fibrosis correctly identified by the Fibrometer test

SECONDARY OUTCOMES:
rate of patients referred to the specialist following the screening procedure, with eLIFT test | 1 day
  Rate of patients with positive screening test (eLIFT ≥8)
rate of patients referred to the specialist following the screening procedure, with FibroMeter test | 1 day
  Rate of patients with positive screening test (FibroMeter ≥0.46)
Rate of "unnecessary referrals" to the specialist with eLIFT test | 1 month
  Rate of patients with positive screening test (eLIFT ≥8) but without final diagnosis of ALF
Rate of "unnecessary referrals" to the specialist with Fibrometer test | 1 month
  Rate of patients with positive screening test (FibroMeter ≥0.46) but without final diagnosis of ALF
Number of hepatocellular carcinoma adetected following the screening procedure, with comparison between eLIFT and FibroMeter strategies | 1 month
  Number of patients with hepatocellular carcinoma (diagnosed on MRI by the recommended radiological criteria: hyperenhancement on the arterial phase and washout on the portal venous phase, or by liver biopsy);
Number of gastroesophageal varices at risk of bleeding detected following the screening procedure, with comparison between eLIFT and FibroMeter strategies | 1 month
  Number of patients with gastroesophageal varices at risk of bleeding (diagnosed by upper-gastrointestinal endoscopy: medium-large varices or small varices with red wall marks)
directs costs by type of disease such as ALF, hepatocellular carcinoma, gastroesophageal varices at risk of bleeding with comparison between eLIFT and FibroMeter strategies | 1 month
  Mean direct cost per patient; mean direct cost generated to detect one patient with ALF, one patient with hepatocellular carcinoma, one patient with gastroesophageal varices at risk of bleeding
eLIFT and FibroMeter screening procedures as a function of the cause of the underlying liver disease (NAFLD, ALD, or mixed NAFLD+ALD) | 1 month
  Rate of patient with ALF, positive screening test, hepatocellular carcinoma, gastroesophageal varices at risk of bleeding, and mean cost, with comparison between NAFLD, ALD, and mixed NAFLD+ALD subgroups
the accuracy of a sequential strategy using eLIFT as first-line test and FibroMeter as second-line test | 1 day
  Rate of patients with ALF diagnosed by a stepwise algorithm using eLIFT ≥8 then, if positive, FibroMeter ≥0.46
patient adherence to the screening of advanced liver fibrosis | 1 month
  Rate of patients included in the study who did not achieve the required screening procedures
most relevant risk factor of advanced liver fibrosis in patients with NAFLD and/or ALD from primary care | 1 day
  Risk factors among clinical characteristics, alcohol consumption, metabolic parameters independently associated with ALF diagnosis
specialized blood test ELF for the screening of advanced liver fibrosis in patients with NAFLD and/or ALD from primary care centers | 1 day
  Same endpoints than primary and secondaries 1 to 11, but using the recommended 9.8 threshold for ELF
Camden and Islington pathway (FIB4 then ELF) for the screening of advanced liver fibrosis in patients with NAFLD and/or ALD from primary care centers, | 1 day
  Same endpoints than primary and secondaries 1 to 11, but using using the Camden and Islington pathway
Camden and Islington pathway , with comparison of sequential strategy eLIFT then FibroMeter | 1 day
  Same endpoints than primary and secondaries 1 to 11, but using using the Camden and Islington pathway

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - ANGERS, Angers
  - CHU Angers, Angers
  - BECON, Bécon-les-Granits
  - Chalonnes, Chalonnes-sur-Loire
  - COMBOURG, Combourg
  - LIFFRE, Liffré
  - Montreuil, Montreuil-Bellay
  - RENNES - Armagnac, Churchill, Rennes
  - RENNES - Kennedy, Rennes
  - CHU Rennes, Rennes
  - SEGRE, Segré
  - Val Couesnon, Val-Couesnon

IPD SHARING:
Plan to Share IPD: No